CLINICAL TRIAL: NCT01569087
Title: Randomized Multicenter Open-label Phase II Clinical Study Comparing the Efficacy and Safety of the Single Dose of Extimia® Versus Daily Filgrastim for Neutropenia Prophylaxis in Breast Cancer Patients Receiving Myelosuppressive Chemotherapy
Brief Title: Dose-finding Study of Empegfilgrastim for Neutropenia Prophylaxis in Patients With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BCD-017-2
Record Dates: First submitted 2012-03-30; First posted 2012-04-02 (Estimated); Results first posted 2016-10-24 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-10

CONDITIONS: Chemotherapy-induced Neutropenia
Keywords: empegfilgrastim; pegylated filgrastim; neutropenia; febrile neutropenia; chemotherapy-associated neutropenia; breast cancer; docetaxel; doxorubicin
MeSH Terms: conditions — Neutropenia; Febrile Neutropenia; Breast Neoplasms | interventions — Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Empegfilgrastim 3 mg (Experimental): Patients will receive a single administration of empegfilgrastim at a dose of 3 mg subcutaneously , 24 h after the chemotherapy
  Interventions: Biological: empegfilrastim
- Empegfilgrastim 6 mg (Experimental): Patients will receive a single administration of empegfilgrastim at a dose of 6 mg subcutaneously, 24 h after the chemotherapy
  Interventions: Biological: empegfilrastim
- Filgrastim (Active Comparator): Patients will receive filgrastim subcutaneously daily (until ANC 10 000/μL or for 14 days, whichever occurred first), starting 24 h after the chemotherapy
  Interventions: Biological: filgrastim

INTERVENTIONS:
Biological: empegfilrastim — Empegfilgrastim is supplied as solution for injection 3 mg/ml. Empegfilgrastim is to be administered 24 h after the chemotherapy at dose of 3 or 6 mg.
  Other Names: Extimia; BCD-017; metpegfilgrastim; pegylated filgrastim; peg-GCSF; empegfilgrastim
  Arms: Empegfilgrastim 3 mg; Empegfilgrastim 6 mg
Biological: filgrastim — Filgrastim should be administered no earlier than 24 hours after the administration of cytotoxic chemotherapy. Filgrastim should be administered daily for up to 2 weeks until the ANC has reached 10 000/mm3 following the expected chemotherapy-induced neutrophil nadir.
  Other Names: GCSF
  Arms: Filgrastim

SUMMARY:
The purpose of the study is to compare safety and efficacy of a single dose of empegfilgrastimt a dose of 3 or 6 mg versus daily administration of filgrastim at a dose of 5 μg/kg/day.

DETAILED DESCRIPTION:
BCD-017-2 is an open-label randomized phase II clinical study to compare the incidence of CTCAE grade 3/4 neutropenia after a single administration of recombinant human pegylated filgrastim empegfilgrastim (Extimia®) at a dose of 3 or 6 mg versus daily administration of filgrastim at a dose of 5 μg/kg/day for neutropenia prophylaxis in breast cancer patients receiving myelosuppressive chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form;
* Histologically verified diagnosis of stage IIb/III/IV breast cancer;
* Age of 18-70 years inclusive;
* If the patient had received the chemotherapy for breast cancer, it should be finished 30 days before the beginning of the study;
* ECOG Performance Status of 0, 1 or 2, not increasing within during 2 weeks before randomization;
* ANC level of 1500/μL and more at the beginning of the study
* Platelet count of 100 000/μL and more at the beginning of the study
* Hemoglobin level of 90 g/l and more
* Creatinine level <1.5 mg/dl
* Total bilirubin level <1.5 × the upper limit of normal (ULN)
* ALT and/or AST levels <2.5×ULN (5×ULN for patients with liver metastases);
* Alkaline phosphatase <5×ULN;
* Left ventricular ejection fraction >50% and more;
* If the patient had received adjuvant and/or neoadjuvant therapy, the cumulative dose of anthracyclines should not exceed 500 mg/m2 for doxorubicin or 500 mg/m2 for epirubicin;
* Ability of the participant to follow the protocol requirements, according to the Investigator's opinion;
* Patients of childbearing potential must implement reliable contraceptive measures during the study treatment, starting 4 weeks prior randomization and for 6 months after the last administration of the study drug.

Exclusion Criteria:

* Patient has received two or more chemotherapy regimens for the metastatic breast cancer;
* Documented hypersensitivity to filgrastim, pegfilgrastim, docetaxel, doxorubicin, dexamethasone and/or its excipients, PEGylated drugs, recombinant proteins.
* Pregnancy or breastfeeding;
* Systemic antibiotic therapy within 72 h prior empegfilgrastim/filgrastim administration;
* Concomitant radiotherapy (except selective radiotherapy of bone metastases);
* Surgery, radiotherapy (except selective radiotherapy of bone metastases), administration of any experimental drugs within 30 days prior randomization;
* History of bone marrow/stem cell transplantation;
* Conditions limiting the patient's ability to follow the protocol;
* CTCAE grade 2/4 neuropathy
* HIV, HCV, HBV, T.Pallidum infection(s);
* Acute or active chronic infections.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-05; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roman A. Ivanov, MD, PhD, Study Director — Biocad
Locations (5):
- Russia (5):
  - Arkhangelsk District Clinical Oncology Dispensary, Arkhangelsk
  - Perm Region Oncology Dispensary, Perm
  - N.N.Petrov Oncology Research Center, Saint Petersburg
  - Russian scientific center of radiology and surgery technologies, Saint Petersburg
  - Volgograd District Oncology Dispensary №1, Volgograd

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Empegfilgrastim 3 mg | Empegfilgrastim 6 mg | Filgrastim
Started | 21 | 20 | 19
Completed | 20 | 20 | 18
Not Completed | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Empegfilgrastim 3 mg | Empegfilgrastim 6 mg | Filgrastim | Total
Number analyzed (Participants) | 21 | 20 | 19 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 20 | 19 | 60
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54.0 [45.9 to 58.8] | 53.5 [48.6 to 57.7] | 48.7 [46.3 to 54.8] | 53.5 [46.5 to 57.1]
Gender [Count of Participants; unit: Participants]
  Female | 21 | 20 | 19 | 60
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russian Federation | 21 | 20 | 19 | 60
Duration of a disease [Median (Inter-Quartile Range); unit: months] | 0.8 [0.4 to 5.8] | 0.6 [0.3 to 2.5] | 0.5 [0.2 to 1.0] | 0.65 [0.33 to 1.58]
Histologic type of a breast cancer [Number; unit: participants]
  ductal | 15 | 11 | 15 | 41
  lobular | 0 | 3 | 0 | 3
  ductal/lobular | 1 | 0 | 0 | 1
  medullar | 2 | 0 | 0 | 2
  no data | 3 | 6 | 4 | 13
Expression of hormone receptors [Number; unit: participants]
  estrogen receptors | 4 | 0 | 2 | 6
  estrogen and progesterone receptors | 7 | 10 | 7 | 24
  deficiency estrogen and progesterone receptors | 9 | 9 | 9 | 27
  no data | 1 | 1 | 1 | 3
HER2 expression [Number; unit: participants]
  1+ | 6 | 3 | 3 | 12
  2+ | 3 | 4 | 3 | 10
  3+ | 6 | 3 | 8 | 17
  deficiency HER2 expression | 5 | 9 | 5 | 19
  no data | 1 | 1 | 0 | 2
History previous therapy of breast cancer [Number; unit: participants]
  yes | 5 | 5 | 4 | 14
  no | 16 | 15 | 15 | 46

OUTCOME MEASURES:

1. Primary Outcome: CTCAE Grade 3/4 Neutropenia Incidence
Time Frame: 21 days
Population: Modified intention-to-treat population (analysis included patients who received at least 1 injection of study drug. Patients who had missed blood sampling on visit 5 [expected time of nadir] were excluded from analysis)
Measure: Number; unit: participants
Arm/Group | Empegfilgrastim 3 mg | Empegfilgrastim 6 mg | Filgrastim
Number analyzed (Participants) | 21 | 20 | 18
participants | 18 | 13 | 11
Statistical Analysis 1: Comparison: Empegfilgrastim 3 mg vs Empegfilgrastim 6 mg vs Filgrastim; Test type: Superiority or Other; p < 0.05, Fisher Exact

2. Secondary Outcome: Mean Duration of CTCAE Grade 4 Neutropenia
Time Frame: 21 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Empegfilgrastim 3 mg | Empegfilgrastim 6 mg | Filgrastim
Number analyzed (Participants) | 21 | 20 | 18
days | 0.43 (0.50) | 0.40 (0.49) | 0.33 (0.47)

3. Secondary Outcome: The Duration of Any Grade Neutropenia
Time Frame: 21 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Empegfilgrastim 3 mg | Empegfilgrastim 6 mg | Filgrastim
Number analyzed (Participants) | 21 | 20 | 18
days | 1.86 (1.39) | 1.0 (0.79) | 0.78 (0.43)

4. Secondary Outcome: Low Level (Nadir) ANC x 10^9/L
Time Frame: 21 days
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: cells x 10^9/L
Arm/Group | Empegfilgrastim 3 mg | Empegfilgrastim 6 mg | Filgrastim
Number analyzed (Participants) | 21 | 20 | 18
cells x 10^9/L | 0.57 [0.3 to 0.73] | 0.75 [0.28 to 1.32] | 0.82 [0.4 to 1.89]

5. Secondary Outcome: Duration of Neutropenia From Nadir to ANC < 2,0 x 10^9 Cells/L on the First Cycle of Chemotherapy
Time Frame: 21 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Empegfilgrastim 3 mg | Empegfilgrastim 6 mg | Filgrastim
Number analyzed (Participants) | 21 | 20 | 18
days | 4.8 (1.64) | 3.8 (2.04) | 3.00 (1.71)

6. Secondary Outcome: Incidence of Febrile Neutropenia
Time Frame: 21 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Empegfilgrastim 3 mg | Empegfilgrastim 6 mg | Filgrastim
Number analyzed (Participants) | 21 | 20 | 18
participants | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Empegfilgrastim 3 mg | Empegfilgrastim 6 mg | Filgrastim
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20 | 2/19
Other Adverse Events (participants affected / at risk) | 21/21 | 20/20 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Empegfilgrastim 3 mg (N=21) | Empegfilgrastim 6 mg (N=20) | Filgrastim (N=19)
neutropenia grade 4 (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Empegfilgrastim 3 mg (N=21) | Empegfilgrastim 6 mg (N=20) | Filgrastim (N=19)
neutropenia grade 3 (Blood and lymphatic system disorders) | 9 (9) | 6 (6) | 6 (6)
neutropenia grade 4 (Blood and lymphatic system disorders) | 9 (9) | 9 (9) | 7 (7)
anemia (Blood and lymphatic system disorders) | 12 (12) | 12 (12) | 15 (15)
white blood cells decreased (Blood and lymphatic system disorders) | 21 (21) | 19 (19) | 17 (17)
Trombocitopenia (Blood and lymphatic system disorders) | 11 (11) | 12 (12) | 6 (6)
febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
hiperglicemia (Endocrine disorders) | 15 (15) | 16 (16) | 16 (16)
ALT decreased (Hepatobiliary disorders) | 8 (8) | 6 (6) | 5 (5)
Alcaline Phosphotase decreased (Hepatobiliary disorders) | 2 (2) | 2 (2) | 6 (6)
alopecia (General disorders) | 8 (8) | 11 (11) | 12 (12)
nousea (General disorders) | 3 (3) | 7 (7) | 5 (5)
fatigue (General disorders) | 7 (7) | 8 (8) | 7 (7)
ossalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 3 (3)
arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
headache (General disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes